CLINICAL TRIAL: NCT05164471
Title: A Dose Confirmation Study of FLT180a (Adeno-associated Viral Vector Containing the Padua Variant of a Codon-optimized Human Factor IX Gene) in Adult Subjects With Hemophilia B
Brief Title: Phase 1/2 Dose Confirmation Study of FLT180a in Hemophilia B
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Freeline has decided to pause development of FLT180a for business priorities
Sponsor: Spur Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FLT180a-06
Record Dates: First submitted 2021-11-22; First posted 2021-12-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FLT180a (Experimental): A single dose of FLT180a will be administered. Dose will be determined by enrollment cohort. The first 3 patients will receive 7.7 x 10e11 vg/kg. The dose in subsequent cohorts will be determined by the DMC based on review of data from the prior cohort(s).
  Interventions: Genetic: verbrinacogene setparvovec

INTERVENTIONS:
Genetic: verbrinacogene setparvovec — FLT180a is a gene therapy intended to increase endogenous FIX production in adults with Hemophilia B

SUMMARY:
Study of FLT180a gene therapy in adults with Hemophilia B. Up to 9 patients will be enrolled to receive a single dose of FLT180a and be followed for 52 weeks. Results will confirm the dose for a future Phase 3 study.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of Hemophilia B with known severe or moderately severe FIX deficiency (≤2% normal circulating FIX activity) for which the subject is on continuous, stable and adequate FIX prophylaxis
* Have acceptable laboratory values of a) Hemoglobin ≥11g/dL; b) Platelets ≥100,000 cells/µL; c) AST, ALT and alkaline phosphatase (ALP) ≤ upper limit of normal (ULN); d) Serum albumin > lower limit of normal (LLN); e) Total bilirubin ≤1.5 x ULN (except if caused by Gilbert's disease); f) Serum creatinine ≤2.0mg/dL.
* Level of neutralizing anti-AAV-S3 antibodies below the limit of the pre-established clinical cutoff using an in vitro transduction inhibition assay within the 4 weeks prior to FLT180a administration
* Has demonstrated ability to accurately, independently and in a timely manner enter bleed diary data during the lead-in study, as judged by the investigator
* At least 150 exposure days to FIX concentrates
* At least 6 months of satisfactory controlled prospective baseline data for bleeding events and FIX consumption data from the FLT-01 lead-in study (ECLIPSE)

Key Exclusion Criteria:

* Any history of alcohol or drug dependence
* Presence of neutralizing anti human FIX antibodies (inhibitor; determined by the Nijmegen modified Bethesda inhibitor assay) at the time of enrolment or a previous history of FIX inhibitor
* Subjects at high risk of thromboembolic events
* Evidence of advanced liver fibrosis
* Prior treatment with a gene transfer medicinal product
* Subjects with active hepatitis B or C
* Serological evidence of HIV-1, not controlled with anti-viral therapy and as evidenced by cluster of differentiation 4 (CD4)+ counts ≤200 μL
* Cytomegalovirus (CMV) immunoglobulin G positive subjects who are CMV polymerase chain reaction (PCR) positive at screening
* Known coagulation disorder other than hemophilia B
* High sensitivity (hs) troponin-T ≥14 pg/mL during screening
* History of uncontrolled cardiac failure, unstable angina, or myocardial infarction or other acute cardiac conditions requiring clinical management in the past 6 months
* Planned surgical procedure within the next 12 months requiring prophylactic FIX treatment
* Known active severe infection (including documented coronavirus (COVID)-19 infection), or any other significant concurrent, uncontrolled medical condition

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of FLT180a as assessed by incidence and severity of AEs and SAEs | Post-dose through week 52
Assessment of FIX activity levels to allow dose confirmation for future Phase 3 study | Assessment at Day 21 post-dose
Assessment of FIX activity levels to allow dose confirmation for future Phase 3 study | Assessment at Day 140 post-dose
Assessment of FIX activity levels to allow dose confirmation for future Phase 3 study | Assessment at Day 182 post-dose

SECONDARY OUTCOMES:
Assessment of change in annualized bleeding rate (ABR) | Pre-dose and Week 52 post-dose
Assessment of change in annualized FIX concentrate consumption | Pre-dose and Week 52 post-dose
Proportion of subjects achieving FIX activity level above 40% | Week 26
The proportion of subjects remaining free from continuous routine FIX prophylaxis | Post dose through week 52
The proportion of subjects achieving a FIX activity level between 50-150% | Pre-dose and Week 52
Assessment of health-related Quality of Life Questionnaire (measuring physical health, feelings, sport and leisure, dealing with haemophilia treatment) (Haem-A-QoL questionnaire) | Pre-dose and Weeks 26, 52 post-dose
Joint bleeding rates | Pre-dose and Week 52
Spontaneous bleeding rates | Pre-dose and Week 52
Number of target joints | Pre-dose and Week 52
Assessment of Quality of Life Questionnaire (measuring mobility, self-care, usual activities, pain/discomfort & anxiety/depression)(EQ-5D-5L questionnaire). | Pre-dose and Weeks 26, 52 post-dose
Measurement of Anti-AAVS3 antibodies and neutralizing antibodies | Pre-dose, Week 4 and Week 26
Evaluation of AAVS3 capsid-specific T-cell reactions | Pre-dose, Week 4 and Week 26
Abnormal or change from baseline findings for liver ultrasound | Pre-dose and Week 52
Abnormal or change from baseline findings for serum alpha-fetoprotein (AFP) levels. | Pre-dose and Week 52
FIX inhibitor level | Pre-dose through Week 52
Use of immunosuppressants (dose and duration per participant) for the prevention and treatment of increased Liver Enzymes | Pre-dose through Week 52
Clearance of vector genomes in plasma and semen as assessed by PCR test | Pre-dose through Week 52
Assessment of Clinically significant changes in 12-lead ECG | Pre-dose through Week 26

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of South Florida, Tampa, Florida
  - University of Michigan, Ann Arbor, Michigan
- United Kingdom (4):
  - Glasgow Royal Infirmary, Glasgow
  - Guys Hospital, London
  - Royal Free London NHS Foundation Tust, London
  - Royal Victoria Infirmary, Newcastle

IPD SHARING:
Plan to Share IPD: No